CLINICAL TRIAL: NCT06779136
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study Evaluating the Efficacy and Safety of a Humanized MG-K10 Mab Injection in Subjects With Prurigo Nodularis.
Brief Title: Phase III Clinical Study of MG-K10 Humanized Mab Injection in Subjects With Prurigo Nodularis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-K10-PN-001
Record Dates: First submitted 2024-12-30; First posted 2025-01-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo nodularis

STUDY DESIGN:
Intervention Model Description: A phase III clinical study to evaluate the efficacy and safety of a humanized MG-K10 mab injection in subjects with prurigo nodularis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MG-K10 Humanized Monoclonal Antibody Injection (Experimental): Every four weeks, subcutaneous injection ，total of 56W
  Interventions: Drug: Placebo
- placebo (Placebo Comparator): Every four weeks, subcutaneous injection，Switch to MG-K10 treatment after 24 weeks of administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Every four weeks, subcutaneous injection，Switch to MG-K10 treatment after 24 weeks of administration

SUMMARY:
A phase III clinical study to evaluate the efficacy and safety of a humanized MG-K10 mab injection in subjects with prurigo nodularis.administered every 4 weeks for 56 weeks.

DETAILED DESCRIPTION:
The study was a multicenter, randomized, double-blind, placebo-controlled Phase III study. Approximately 160 adults with prurigo nodularis were scheduled to receive multiple subcutaneous injections (every 4 weeks for 56 weeks). The study was divided into a screening period (1-4 weeks), a double-blind treatment period (24 weeks), a maintenance treatment period (24 weeks), and a follow-up period (8 weeks).

ELIGIBILITY:
eligibility criteria:

1. voluntarily sign the ICF and comply with all the visits and research-related procedures required by the protocol;
2. Both men and women were required to be ≥ 18 and ≤ 80 years old at the time of signing the informed consent;
3. the duration of PN diagnosed by a dermatologist at the time of screening was ≥ 3 months;
4. In the range of 1-10, WI-NRS≥7 in the past 24 h at screening; WI-NRS in the week before the baseline visit The average weekly score was ≥ 7 points.

Exclusion criteria：

1. There are skin diseases other than PN and mild atopic dermatitis (AD) that may interfere with the assessment of research outcomes.
2. Patients who had a history of moderate to severe AD during the 6 months prior to the screening visit or screening visit.
3. Receiving potent or super-potent TCS/TCI treatment within 2 weeks before or during screening.

4) Evidence of active tuberculosis. 5) Participation in any other clinical study within 12 weeks or 5 half-lives prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportions of subjects achieving WI-NRS | week 24
  In the experimental group, the weekly mean value of WI-NRS at week 24 was compared with baseline.Proportion of subjects who improved (decreased) by ≥ 4 points

SECONDARY OUTCOMES:
Proportions of subjects achieving IGA PN-S score of 0/1 point | week 24
  Proportion of subjects with overall disease score of 0/1
The proportion of subjects whose weekly mean WI-NRS decreased by ≥ 4 from baseline at each evaluation visit | From baseline to week 56
  The proportion of subjects whose weekly mean WI-NRS decreased by ≥ 4 from baseline at each evaluation visit
The absolute value and percentage change of weekly mean WI-NRS from baseline at each evaluation visit; | From baseline to week 56
  The absolute value and percentage change of weekly mean WI-NRS from baseline at each evaluation visit;
Duration of onset of response to pruritus | From baseline to week 56
  The proportion of subjects with a weekly mean decrease of ≥4 points from baseline in the WI-NRS was compared, and the difference from the placebo group was first presented p < 0.05).
the first response to pruritus occurred. | from baseline to the week 24
  The time from baseline to the 24th week when the first response to pruritus occurred (the average weekly WI-NRS score decreased by ≥ 4 points compared with the baseline)
The time when the first intergroup response difference in pruritus occurred | From baseline to week 24
  The time of the first intergroup response difference for pruritus (the time when the difference in the proportion of subjects with a weekly average WI-NRS score reduction of ≥ 4 points compared to the baseline first reached p < 0.05 compared with the placebo group)
The duration of the difference in persistent response to pruritus between groups | From baseline to week 24
  The duration of the difference in persistent response between the prurity-onset groups (comparing the change in weekly WI-NRS from baseline between the MG-K10 and placebo groups, the time when the difference between the MG-K10 and placebo groups first appeared to be p < 0.05 and remained significant on subsequent measures)
Proportion of subjects with an IGA PN-S score of 0/1 | From baseline to week 56
  Proportion of subjects with IGA PN-S score of 0/1 at each evaluation visit
Changes in IGA PN-S scores | From baseline to week 56
  Changes in IGA PN-S scores from baseline at each evaluation site
Proportion of subjects with an IGA PN-A score of 0/1 | From baseline to week 56
  Proportion of subjects with an IGA PN-A score of 0/1 from baseline to each visit point
Changes in IGA PN-A scores from baseline | From baseline to week 56
  Changes in IGA PN-A scores from baseline at each evaluation visit
Proportion of subjects wit weekly WI-NRS improvement (decrease) of ≥ 4 points and IGA PN-S of 0/1 | From baseline to week 56
  Proportion of subjects with weekly WI-NRS improvement (decrease) of ≥ 4 points from baseline and IGA PN-S of 0/1 at each evaluation visit
Changes in DLQI scores from baseline | From baseline to week 56
  Change in Dermatology Life Quality Index (DLQI) from baseline at each evaluation visit
Changes in HADS from baseline | From baseline to week 56
  Changes in Hospital Anxiety and Depression Scale(HADS) from baseline at each evaluation site
safety | From baseline to week 56
  These include Treatment Emergent Adverse Events (TEAE) and Serious Adverse events Events (SAE), adverse events of special interest (AESI), clinical laboratory tests, vital signs, physical examination, and abnormalities in 12-lead electrocardiograms;
pharmacokinetics | From baseline to week 56
  Ctrough (valley concentration) change over time;
pharmacodynamics | From baseline to week 56
  Changes of biomarkers before and after administration
immunogenicity | From baseline to week 56
  Occurrence of Anit-Drug Antibodies (ADA) and Neutralizing Antibodies (NAb)

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Medical Ph.D, Study Director — Feking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing,, Beijing, Bejing, China

IPD SHARING:
Plan to Share IPD: No